CLINICAL TRIAL: NCT00775424
Title: A PHASE Ib PARTIALLY RANDOMIZED PILOT STUDY INTENDED TO EVALUATE THE SAFETY AND IMMUNOLOGICAL EFFECTS OF HIV-1 DNA IMMUNIZATION (PENNVAX-B) WITH OR WITHOUT CO-ADMINISTRATION OF CONSTRUCTS CONTAINING DNA ENCODING FOR THE EXPRESSION OF EITHER IL-12 OR IL-15 IN HIV INFECTED INDIVIDUALS
Brief Title: PENNVAX-B With or Without IL-12 or IL-15 as a DNA Vaccine for HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807682
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: HIV Infection
Keywords: HIV infection; DNA vaccine; IL-12 adjuvant; IL-15 adjuvant
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PENNVAX-B alone (Experimental): PENNVAX-B alone
  Interventions: Biological: PENNVAX-B
- PENNVAX-B+IL12 (Experimental): PENNVAX-B+IL12
  Interventions: Biological: PENNVAX-B; Biological: GENEVAX IL-12-4532
- PENNVAX-B+IL15 (Experimental): PENNVAX-B+IL15
  Interventions: Biological: PENNVAX-B; Biological: IL-15 adjuvant
- PLACEBO (Placebo Comparator): PLACEBO
  Interventions: Biological: PLACEBO

INTERVENTIONS:
Biological: PENNVAX-B — PENNVAX-B is a cocktail of three expression plasmids. The plasmids include the genes which encode a synthetic HIV-1 envelope protein (pEY2E1-B), Gag (gagCAM02), and Pol (pK2C1). Each plasmid is manufactured to a concentration of 4.0 mg/mL and is formulated with bupivacaine (0.25%) as a facilitating agent for DNA uptake. All plasmids (2.0 mg each gag, pol, env) are premixed by the manufacturer in the same vial.
  Arms: PENNVAX-B alone; PENNVAX-B+IL12; PENNVAX-B+IL15
Biological: GENEVAX IL-12-4532 — GENEVAX IL-12-4532 This molecular adjuvant plasmid contains nucleotide sequences necessary for expression of the human IL-12 protein. IL-12 DNA is formulated at a concentration of 2.0 mg/mL with bupivacaine (0.25%).
  Arms: PENNVAX-B+IL12
Biological: PLACEBO — PLACEBO
  Arms: PLACEBO
Biological: IL-15 adjuvant — pIL15EAM is a plasmid that encodes human IL-15 and has been optimized to express 87 fold higher than native IL-15 DNA and 5.7 fold higher than an earlier generation optimized IL-15 DNA construct. This plasmid is formulated at a concentration of 4.0 mg/mL with bupivacaine (0.25%).
  Arms: PENNVAX-B+IL15

SUMMARY:
A phase Ib partially blinded pilot study to evaluate the safety and immunological effects of PENNVAX-B with or without co-administration of constructs containing DNA encoding for the expression of either IL-12 or IL-15.

Primary objectives

1. To determine the safety of HIV-1 DNA constructs (PENNVAX-B).
2. To determine the safety and optimal doses of the IL-12 and the IL-15 adjuvant constructs when given with PENNVAX-B.

Secondary objectives

1. To compare the various vaccine groups for their immunological responses to several HIV-1 antigens, utilizing the ELISPOT assay.
2. To analyze antibody responses to the vaccine antigens over time.
3. To measure CD8 cell proliferative responses to vaccine antigens over time.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection documented by any licensed ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, or plasma HIV-1 RNA, at any time before study entry.
2. Taking a stable HAART regimen for ≥3 months before the time of enrollment.
3. CD4-positive lymphocyte count ≥400 cells/µl on two occasions within 60 days of enrollment, performed at any certified flow laboratory.
4. HIV-1 < 75 copies/mL on two occasions within 60 days of enrollment, performed in a CLIA certified laboratory.
5. Laboratory values obtained within 30 days prior to study entry:
6. Hemoglobin > 9 g/dL (female subjects) and > 9.5 g/dL (male subjects)
7. Absolute neutrophil count > 1000 cells/μL
8. Platelet count > 75,000/μL
9. ALT, AST and alkaline phosphatase ≥ 2.5 x upper limit of normal range
10. Total bilirubin ≥ 2.5 x upper limit of the laboratory normal range
11. Serum creatinine ≥ upper limit of normal (ULN).
12. All women of reproductive potential (who have not reached menopause nor undergone hysterectomy, oophorectomy, or tubal ligation) must have a negative pregnancy test within 30 days of initiating study-specified medication(s) and at day 0 (enrollment).

    1. Women who are not of reproductive potential (have reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation) or whose male partner has undergone successful vasectomy with resultant azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Documentation of menopause, sterilization (hysterectomy, oophorectomy, tubal ligation, or vasectomy) and azoospermia by patient-reported history is acceptable.
    2. All subjects must not participate in a conception process (i.e. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use a form of contraception while receiving protocol-specified medication(s)/vaccinations and for one month after stopping the vaccinations.
13. Karnofsky performance score ≥ 90 within 30 days prior to study entry.
14. Men or women ≥18 years of age and less than 50.
15. Ability and willingness of subject or legal guardian/representative to give written informed consent.

Exclusion Criteria:

1. Any active or past AIDS-defining illness with the exception of minimal (less than 10 lesions) cutaneous Kaposi's sarcoma.
2. Subjects with a history of a CD4+ T-cell count ≤200/µl are not eligible.
3. Use of any known immunomodulatory therapy within 4 weeks prior to study entry including but not limited to drugs such as systemic corticosteroids, interferons, interleukins, thalidomide, granulocyte-macrophage colony-stimulating factor, IV gammaglobulin, or human growth hormone.
4. Any malignancy requiring systemic or local toxic chemotherapy. Local radiation will be allowed.
5. Pregnancy or breast-feeding.
6. Uncontrolled diabetes mellitus (fasting blood glucose > 126 mg/dL or random blood glucose levels > 200 mg/dL on at least two occasions within 6 months prior to study entry).
7. Major organ transplantation.
8. Active alcohol or substance abuse or psychiatric illness, which in the opinion of the investigator will interfere with adherence to study requirements.
9. Clinically significant neurological disorder occurring within 1 year prior to study entry that in the opinion of the principal investigator would affect the subject's study compliance or safety.
10. Use of systemic corticosteroids for ≥ 4 weeks within 3 months prior to study entry.
11. Presence of any chronic disease that in the opinion of the investigator might affect subject safety.
12. History of previous vaccination with an HIV-1 vaccine.
13. History or evidence of autoimmune disease, including, but not limited to thyroid autoimmune disease and idiopathic thrombocytopenic purpura.
14. Allergies to bupivacaine or similar anesthetic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events in each of the treatment arms | Time of each vaccination, 2 weeks after vaccinations 3 and 4 and at the completion of the study.

SECONDARY OUTCOMES:
Antigen specific cellular and humoral immune response. | 2 weeks following the third and fourth vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania. Clinical Trials Unit, Philadelphia, Pennsylvania, United States